CLINICAL TRIAL: NCT05359939
Title: A Head-to-head Comparison of MRI, CT, 18F-FDGal and 18F-choline in Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-288-20
Record Dates: First submitted 2022-04-19; First posted 2022-05-04 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Head-to-head comparison of two tracers: 18F-FDGal PET/CT, 18F-choline PET/CT (Other): Diagnostic scan
  Interventions: Diagnostic Test: 18F-FDGal PET/CT versus 18F-choline PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDGal PET/CT versus 18F-choline PET/CT — Fifty patients with known HCC are investigated with two PET/CT-scans with 18F-FDGal and 18F-choline. In some of the cases one of the CT-scans will be altered to a contrast-enhanced MRI scan. A contrast-enhanced CT scan will be performed as part of the standard diagnostic work-up. We include patients with known HCC as the aim is to compare the diagnostic performance of the two tracers. Images will be analyzed for focal lesions and compared to other modalities by an experienced specialist in PET and an experienced radiologist.

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver tumour and is the fourth leading cause of cancer-related death worldwide. In Denmark, the incidence of HCC is 5.2 per 100.000 population per year with a dismal prognosis as the median survival time is just 7.7 month. Extrahepatic spread of HCC is common at advanced stages.

The majority of patients who develop HCC has cirrhosis of the liver and in these patients, diagnosis can be made non-invasively with characteristic contrast-enhancement pattern on CT and/or MRI. Although contrast-enhanced CT and MRI are considered equal in current guidelines, MRI may have a better sensitivity especially for small lesions.

Positron emission tomography (PET) is a molecular imaging technique based on the injection of a very small dose of a tracer substance labelled with a positron emitting radioisotope. PET with the glucose tracer 18F-FDG is an important tool in the staging of many cancer forms, but it is not included in the international guidelines for management of HCC because of suboptimal sensitivity of only up to 50-60 % for HCC situated in the liver. Other PET tracers such as 11C- or 18F-choline have also been investigated in patients with HCC with detection rates of 84% in meta-analysis.

In Aarhus, the liver specific tracer 18F-FDGal has been developed. It is a fluorine-18 labelled galactose analogue which in the human body is trapped in hepatocytes by phosphorylation by galactokinase. The first study of the diagnostic use of 18F-FDGal PET/CT in patients suspected for having HCC was published in 2011. The study showed good clinical potential for 18F-FDGal as a tracer for detection of intra- as well as extrahepatic HCC.

Both 18F-choline and 18F-FDGal show potential to improve the detection of extrahepatic disease. Some centres use 18F-choline PET/CT in evaluation of patients with HCC, but the reported results for choline PET/CT do not appear superior to 18F-FDGal PET/CT. Furthermore, 18F-FDGal PET/CT also enables evaluation of regional metabolic liver. A head-to-head study of the two tracers is very much warranted.

The aim of the present project is to establish the clinical impact and utilization of 18F-FDGal PET in concert with state-of-the art radiological methods (CT and MRI) in patients with HCC.

Hypotheses:

i) 18F-FDGal PET performs better than 18F-choline for diagnosis and staging of patients with HCC.

ii) MRI is expected to perform better than contrast-enhanced CT.

ELIGIBILITY:
Inclusion Criteria:

* patients with hepatocellular carcinoma
* age above 18 years

Exclusion Criteria:

* the patient does not want to take part in the study
* the responsible investigator determines that the patient is not qualified for a PET scan
* a history of moderate or intense hypersensitivity to a gadolinium-based contrast agent
* renal insufficiency (estimated glomerular filtration rate [eGFR] <30 ml/min/1.73 m2 body surface area
* contraindications for MRI including claustrophobia
* pregnant or nursing patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hepatocellular carcinoma - sensitivity and specificity of two PET tracers | Three years
  The ability of the scans 18F-FDGal PET/CT or PET/MRI and 18F-choline PET/CT or PET/MRI to correctly identify lesions representing intrahepatic and/or extrahepatic hepatocellular carcinoma.

SECONDARY OUTCOMES:
Hepatocellular carcinoma - sensitivity and specificity of MRI and CT | Three years
  The ability of MRI and CT to correctly identify lesions representing hepatocellular carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
According to local rules and GDPR it is not possible for study data to leave the facility.